CLINICAL TRIAL: NCT00070109
Title: A Phase II Study Of Trabectedin (ET-743, Yondelis®) in Children With Recurrent Rhabdomyosarcoma, Ewing Sarcoma, or Nonrhabdomyosarcomatous Soft Tissue Sarcomas
Brief Title: Trabectedin in Treating Young Patients With Recurrent or Refractory Soft Tissue Sarcoma or Ewing's Family of Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0221; NCI-2009-00357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000329999 (Other: Clinical Trials.gov); COG-ADVL0221 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma; Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Trabectedin 1.3 mg/m2 to assess feasibility in all patients (Experimental): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity. A cohort of 6 patients will be enrolled at the 1.3 mg/m2 dose level.
  Interventions: Drug: trabectedin; Other: pharmacological study
- Trabectedin 1.5 mg/m2 to assess feasibility in all patients (Experimental): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity. Six toxicity-evaluable patients are assigned this treatment.
  Interventions: Drug: trabectedin; Other: pharmacological study
- Trabectedin at 1.5 mg/m2 to assess efficacy in Ewing sarcoma (Experimental): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: trabectedin; Other: pharmacological study
- Trabectedin at 1.5 mg/m2 - assess efficacy in rhabdomyosarcoma (Experimental): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: trabectedin; Other: pharmacological study
- Trabectedin 1.5 mg/m2 - assess efficacy in nonrhabdomyosarcoma (Experimental): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: trabectedin; Other: pharmacological study

INTERVENTIONS:
Drug: trabectedin — Given IV
  Other Names: Ecteinascidin; ET 743; Yondelis
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well trabectedin works in treating young patients with recurrent or refractory soft tissue sarcoma or Ewing's family of tumors. Drugs used in chemotherapy such as trabectedin use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in pediatric patients with recurrent or refractory soft tissue sarcomas or Ewing's sarcoma family of tumors treated with ecteinascidin 743 (trabectedin).

II. Determine the toxicity of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients.

OUTLINE:

Patients receive trabectedin IV over 3 hours on day 1. Treatment repeats every 21days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 12 months of age at the time of study entry and no more than 21 years of age when initially diagnosed with the malignancy to be treated on this protocol
* Histologically confirmed recurrent or refractory sarcoma tumors, including the following:

  * Rhabdomyosarcoma
  * Nonrhabdomyosarcomatous soft tissue sarcoma
  * Ewing's sarcoma
* Measurable disease by imaging studies

  * Lesions assessable only by radionuclide scans are not considered measurable
  * If the only measurable lesion has been previously irradiated, then that lesion must have shown evidence of an interim increase in size
* No significant amount of metastatic liver disease, defined as the following:

  * Lesions occupying more than 25% of the liver by imaging and abnormal liver function tests or abnormal synthetic liver function
* Performance status - Lansky 50-100% (10 years of age and under)
* Performance status - Karnofsky 50-100% (over 10 years of age)
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (transfusion allowed)
* No concurrent CYP3A4 inhibitors, including the following:

  * Grapefruit juice
  * Erythromycin
  * Azithromycin
  * Clarithromycin
  * Rifampin and its analogs
  * Fluconazole
  * Ketoconazole
  * Itraconazole
  * Cimetidine
  * Cannabinoids (marijuana or dronabinol)
  * Leukotriene inhibitors used in asthma (e.g., zafirlukast, montelukast, or zileuton)
* Bilirubin no greater than upper limit of normal (ULN)
* Total alkaline phosphatase no greater than ULN
* Hepatic fraction alkaline phosphatase and 5 nucleotidase no greater than ULN
* SGOT and SGPT ≤ 2.5 times ULN
* Albumin ≥ 2.5 g/dL
* Gamma-glutamyl transferase < 2.5 times ULN
* Maximum creatinine based on age as follows:

  * 0.8 mg/dL (5 years of age and under)
  * 1.0 mg/dL (6 to 10 years of age)
  * 1.2 mg/dL (11 to 15 years of age)
  * 1.5 mg/dL (over 15 years of age)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) at least 70 mL/min
* No uncompensated congestive heart failure within the past 6 months
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 2 months after study participation
* No active uncontrolled infection
* Weight ≥ 15 kilograms
* More than 1 week since prior growth factors that support platelet or white blood cell number or function
* At least 7 days since prior biologic agents and recovered
* No prior allogeneic stem cell transplantation
* No other concurrent immunomodulating agents
* More than 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No more than 2 prior multi-agent chemotherapy regimens
* No other concurrent anticancer chemotherapy
* Concurrent steroids allowed
* At least 6 weeks since prior since prior extended radiotherapy and recovered
* No prior total body radiotherapy
* Concurrent radiotherapy to localized painful lesions allowed provided at least 1 measurable lesion is not irradiated*
* At least 7 days since prior enzyme-inducing anticonvulsants (e.g., carbamazepine, phenobarbital, or phenytoin)
* No concurrent enzyme-inducing anticonvulsants
* No other concurrent investigational agents

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Baruchel, MD, Principal Investigator — Children's Oncology Group
Locations (14):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital Central California, Madera, California
  - Childrens Memorial Hospital, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Vermont, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Result] Baruchel S, Pappo A, Krailo M, Baker KS, Wu B, Villaluna D, Lee-Scott M, Adamson PC, Blaney SM. A phase 2 trial of trabectedin in children with recurrent rhabdomyosarcoma, Ewing sarcoma and non-rhabdomyosarcoma soft tissue sarcomas: a report from the Children's Oncology Group. Eur J Cancer. 2012 Mar;48(4):579-85. doi: 10.1016/j.ejca.2011.09.027. Epub 2011 Nov 14. PMID 22088484

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients | Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma
Started | 8 | 6 | 8 | 20 | 8
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 8 | 20 | 8
Not completed — Death | 1 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 6 | 4 | 5 | 15 | 5
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 4 | 2
Not completed — removed from prot thpy prior to chemo | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients: Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  trabectedin: Given IV
  pharmacological study: Correlative studies
- Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients; Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma; Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma; Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma: Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  trabectedin: Given IV
- Total: Total of all reporting groups
Arm/Group | Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients | Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma | Total
Number analyzed (Participants) | 8 | 6 | 8 | 20 | 8 | 50
Age, Continuous [Median (Full Range); unit: years] | 18.5 [8 to 24] | 15.5 [8 to 21] | 16 [8 to 20] | 14.5 [4 to 22] | 16 [8 to 21] | 15.5 [4 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 11 | 2 | 19
  Male | 7 | 4 | 5 | 9 | 6 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 3 | 7
  Not Hispanic or Latino | 8 | 5 | 0 | 16 | 5 | 34
  Unknown or Not Reported | 0 | 0 | 8 | 1 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 5 | 1 | 7
  White | 6 | 6 | 7 | 12 | 7 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 5 | 19 | 8 | 43
  Canada | 3 | 0 | 3 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Response (Complete Response [CR] and Partial Response [PR])
Description: Any patient who is enrolled and receives at least one dose of trabectedin will be considered evaluable for response if the individual receives at least one dose of trabectedin and: (1) is removed from protocol therapy because of progressive disease where progressive disease is documented either by imaging studies or clinical progression; or (2) has at least one radiographic evaluation of disease status after the start of protocol therapy and is not electively removed from protocol therapy with stable disease or is not lost to follow-up with stable disease. Patients who achieve a complete response (CR) - disappearance of all target lesions or partial response (PR) - >=30% decrease in the sum of the longest diameter of target lesions according to the RECIST criteria will be considered responders for the study design. All other patients who are evaluable for response will be considered non-responders for the study.
Time Frame: Twenty-six (26) cycles of chemotherapy or termination of protocol therapy, whichever occurs first.
Population: No pts in Group 1 were evaluated for response. 1 pt in Group 3 is excluded because the pt was removed from protocol therapy after cycle 3 when a cardiac evaluation was missed. The pt was removed prior to disease assessment on protocol therapy. 1 pt enrolled in Group 4 was excluded because patient was removed from therapy prior to chemotherapy.
Measure: Number; unit: participants
Groups:
- Trabectedin 1.5 mg/m2- Feasibility in All Patients(Group 2); Trabectedin 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3); Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4); Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  trabectedin: Given IV
Arm/Group | Trabectedin 1.5 mg/m2- Feasibility in All Patients(Group 2) | Trabectedin 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3) | Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4) | Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5)
Number analyzed (Participants) | 6 | 7 | 19 | 8
participants | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Dose-Limiting Toxicity (DLT)
Description: Any Grade 3 or Grade 4 non-hematologic toxicity attributable to the Investigational drug with the specific exclusion of: Grade 3 nausea and vomiting; Grade 3 transaminase (AST/ALT) elevation that return to less than or equal to Grade 1 or baseline prior to the time for the next treatment cycle; Grade 3 fever or infection; Alopecia; Grade 4 neutropenia of > 7 days duration or Grade 4 thrombocytopenia of > 7 days duration, which requires transfusion therapy on greater than 2 occasions in 7 days, or which causes a delay of more than 14 days beyond the planned interval between treatment cycles.
Time Frame: 1 Cycle
Population: Two pts in Group 1 and 1 pt in Group 2 were excluded because they were removed from therapy prior to the DLT evaluation period and no DLT had been observed. No patients in Groups 3, 4, or 5 were evaluated for DLT.
Measure: Number; unit: participants
Groups:
- Trabectedin 1.3 mg/m2- Feasibility in All Patients (Group 1): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  trabectedin: Given IV
  pharmacological study: Correlative studies
- Trabectedin 1.5 mg/m2- Feasibility in All Patients (Group 2): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity. Six toxicity-evaluable patients are assigned this treatment.
  trabectedin: Given IV
Arm/Group | Trabectedin 1.3 mg/m2- Feasibility in All Patients (Group 1) | Trabectedin 1.5 mg/m2- Feasibility in All Patients (Group 2)
Number analyzed (Participants) | 6 | 5
participants | 1 | 0

3. Primary Outcome: Pharmacokinetics by a Miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method : Maximum Plasma Concentration (Cmax) of Trabectedin
Description: The plasma concentrations at each time point were determined by miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method. The plasma concentration-versus-time data of trabectedin were estimated using non-compartmental methods. Individual time points were not available, so one estimated Cmax was derived for each patient.
Time Frame: From baseline up to168 hours after trabectedin infusion in course 1
Population: Patients for whom specimens were submitted to the pharmacokinetics laboratory with sufficient samples to calculate maximum plasma concentration of trabectedin. Group 1 and group 2 patients were excluded due to not submitting specimens.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trabectedin at 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3); Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4); Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5): Patients receive trabectedin over 3 hours on day 1. Treatment repeats every 21 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Trabectedin at 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3) | Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4) | Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5)
Number analyzed (Participants) | 3 | 2 | 5
ng/mL | 3.643333333 (4.08) | 2.285 (0.191) | 1.889 (1.26)

4. Primary Outcome: Pharmacokinetics by a Miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method : Apparent Volume at Steady State (Vss) of Trabectedin
Description: The plasma concentrations at each time point were determined by miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method. The plasma concentration-versus-time data of trabectedin were estimated using non-compartmental methods. Individual time points were not available, so one estimated Vss was derived for each patient.
Time Frame: From baseline up to168 hours after trabectedin infusion in course 1
Population: Patients for whom specimens were submitted to the pharmacokinetics laboratory with sufficient samples to calculate apparent volume at steady state of trabectedin of trabectedin. Group 1 and group 2 patients were excluded due to not submitting specimens.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Trabectedin at 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3) | Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4) | Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5)
Number analyzed (Participants) | 3 | 2 | 2
L | 1860.666667 (999.9) | 1340.5 (439) | 3269.5 (269.4)

5. Primary Outcome: Pharmacokinetics by a Miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method : Half-life of Trabectedin
Description: The plasma concentrations at each time point were determined by miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method. The plasma concentration-versus-time data of trabectedin were estimated using non-compartmental methods. Individual time points were not available, so one estimated Half-life was derived for each patient.
Time Frame: From baseline up to168 hours after trabectedin infusion in course 1
Population: Patients for whom specimens were submitted to the pharmacokinetics laboratory with sufficient samples to calculate trabectedin half life. Group 1 and group 2 patients were excluded due to not submitting specimens.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Trabectedin at 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3) | Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4) | Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5)
Number analyzed (Participants) | 3 | 2 | 2
hours | 47.4 (17.0) | 49.5 (1.70) | 63.4 (22.4)

6. Primary Outcome: Pharmacokinetics by a Miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method : Area Under the Curve (AUC) of Trabectedin
Description: The plasma concentrations at each time point were determined by miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method. The plasma concentration-versus-time data of trabectedin were estimated using non-compartmental methods. Individual time points were not available, so one estimated AUC was derived for each patient.
Time Frame: From baseline up to168 hours after trabectedin infusion in course 1
Population: Patients for whom specimens were submitted to the pharmacokinetics laboratory with sufficient samples to calculate trabectedin AUC. Group 1 and group 2 patients were excluded due to not submitting specimens.
Measure: Mean (Standard Deviation); unit: ng/(mLxh)
Arm/Group | Trabectedin at 1.5 mg/m2- Efficacy in Ewing Sarcoma (Group 3) | Trabectedin 1.5 mg/m2- Efficacy in Rhabdomyosarcoma (Group 4) | Trabectedin 1.5 mg/m2-efficacy in Nonrhabdomyosarcoma(Group 5)
Number analyzed (Participants) | 3 | 2 | 2
ng/(mLxh) | 184.9 (193) | 75.7 (43.3) | 41.2 (18.7)

7. Primary Outcome: Pharmacokinetics by a Miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method : Clearance of Trabectedin
Description: The plasma concentrations at each time point were determined by miniaturized Liquid Chromatography/Tandem Mass Spectrometry Method. The plasma concentration-versus-time data of trabectedin were estimated using non-compartmental methods. Individual time points were not available, so one estimated Clearance was derived for each patient.
Time Frame: From baseline up to168 hours after trabectedin infusion in course 1
Population: Patients for whom specimens were submitted to the pharmacokinetics laboratory with sufficient samples to calculate trabectedin clearance. Group 1 and group 2 patients were excluded due to not submitting specimens.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma
Number analyzed (Participants) | 3 | 2 | 2
L/hr | 20.5786891 (17.9) | 18.11833775 (3.32) | 63.8304367 (29.7)

ADVERSE EVENTS:
Description: 1 patient in Group 4 was not included in the AE analysis as the patient never received treatment.
Arm/Group | Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients | Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/6 | 1/8 | 5/19 | 3/8
Other Adverse Events (participants affected / at risk) | 6/8 | 4/6 | 6/8 | 15/19 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients (N=8) | Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients (N=6) | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma (N=8) | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma (N=19) | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma (N=8)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 1 | 0 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin 1.3 mg/m2 to Assess Feasibility in All Patients (N=8) | Trabectedin 1.5 mg/m2 to Assess Feasibility in All Patients (N=6) | Trabectedin at 1.5 mg/m2 to Assess Efficacy in Ewing Sarcoma (N=8) | Trabectedin at 1.5 mg/m2 - Assess Efficacy in Rhabdomyosarcoma (N=19) | Trabectedin 1.5 mg/m2 - Assess Efficacy in Nonrhabdomyosarcoma (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 1 | 9 | 3
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 5 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 1 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
CPK increased (Investigations) | 1 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 1
Fever (General disorders) | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 1 | 0 | 0 | 5 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 4 | 2
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 2 | 2 | 10 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 5 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 0
White blood cell decreased (Investigations) | 3 | 1 | 2 | 9 | 2
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.